CLINICAL TRIAL: NCT02655653
Title: A Randomized, Double-blinded Trial Comparing the Efficacy of Tranexamic Acid and Epsilon-aminocaproic Acid in Reducing Bleeding and Transfusions in Cardiac Surgery
Brief Title: Efficacy of Tranexamic Acid and Epsilon-aminocaproic Acid in Reducing Bleeding and Transfusions in Cardiac Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Leff, Chief, Cardiothoracic Anesthesiology, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 08-08-291
Record Dates: First submitted 2015-12-31; First posted 2016-01-14 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | US Export: Yes

ARMS (2):
- Epsilon-aminocaproic acid (EACA) (Experimental): Epsilon-aminocaproic acid administered following anesthetic induction: EACA was administered as a bolus loading dose of 150 mg/ kg followed by a maintenance infusion of 15 mg/ kg /hr.
  Interventions: Drug: Epsilon-aminocaproic acid administered
- Tranexamic acid (TA) (Experimental): Tranexamic Acid administered following induction: TA was administered as a bolus dose of 30 mg /kg followed by a 16 mg/ kg/hour maintenance infusion.
  Interventions: Drug: Tranexamic Acid administered

INTERVENTIONS:
Drug: Epsilon-aminocaproic acid administered — Following anesthetic induction, Epsilon-aminocaproic acid was administered as a bolus loading dose of 150 mg/ kg followed by a maintenance infusion of 15 mg/ kg /hr. Maintenance infusion of both drugs was discontinued when the patient arrived in the cardiac surgical intensive care unit. In addition to routine blood sampling ( standard of care in our hospital), patients had thromboelastogram(TEG) and D-dimer levels drawn at the following time points: post incision but prior to initial antifibrinolytic load, immediately following the antifibrinolytic loading dose, and post-protamine reversal of heparin.
  Arms: Epsilon-aminocaproic acid (EACA)
Drug: Tranexamic Acid administered — Following anesthetic induction, Tranexamic Acid was administered as a bolus dose of 30 mg /kg followed by a 16 mg/ kg/hour maintenance infusion. Maintenance infusion of both drugs was discontinued when the patient arrived in the cardiac surgical intensive care unit. In addition to routine blood sampling ( standard of care in our hospital), patients had thromboelastogram(TEG) and D-dimer levels drawn at the following time points: post incision but prior to initial antifibrinolytic load, immediately following the antifibrinolytic loading dose, and post-protamine reversal of heparin.
  Arms: Tranexamic acid (TA)

SUMMARY:
The investigators primary objective is to compare the effectiveness of epsilon-aminocaproic acid (EACA) and tranexamic acid (TA) in reducing bleeding and transfusion in cardiac surgery, with the hypothesis that TA is more effective. The investigators also seek to further examine the clinical benefits and adverse effects profiles of epsilon-aminocaproic acid and tranexamic acid.

DETAILED DESCRIPTION:
This is a single center double blinded randomized controlled study comparing the effectiveness of epsilon-aminocaproic acid (EACA) and tranexamic acid (TA) in reducing 24hour blood transfusion and chest tube drainage. From October 2008 to September 2011, patients greater than 18 years of age, scheduled for cardiac surgery requiring CPB were consented. Eligible operations included; coronary artery bypass graft surgery (CABG), a heart valve repair/replacement, or a concomitant CABG and valve surgery were enrolled.

Consented patients were randomized into one of the two groups using a 1:1 randomization sequence generated by a computer program. Randomization sequence and the study drugs were kept in a locked box and were opened only by unblinded study personnel who were not involved in the clinical care of the patient. This person prepared the study drug following the instructions of the study protocol, resulting in preparations of EACA and TA that contained equi-potent similar volumes of the drug in the syringe, in order to ensure blinding. Antifibrinolytic study drug was administered following anesthetic induction. EACA was administered as a bolus loading dose of 150 mg/ kg followed by a maintenance infusion of 15 mg/ kg /hr. TA was administered as a bolus dose of 30 mg /kg followed by a 16 mg/ kg/hour maintenance infusion. Maintenance infusion of both drugs was discontinued when the patient arrived in the cardiac surgical intensive care unit. In addition to routine blood sampling ( standard of care in the investigators hospital), patients had thromboelastogram(TEG) and D-dimer levels drawn at the following time points: post incision but prior to initial antifibrinolytic load, immediately following the antifibrinolytic loading dose, and post-protamine reversal of heparin.

The primary endpoint was the amount of chest tube drainage and the amount of blood products used in the first 24 hours following surgery (surrogate measurement for blood loss) was measured at 4, 8, 12 and 24 hours after surgery. The incidence of packed red blood cells (PRBC), fresh frozen plasma (FFP), cryoprecipitate and platelets administered during the first 24 hours after surgery was collected. Additionally, patients were monitored for any complications during their stay in the hospital and up to 30 days post-operatively. Complications included renal dysfunction (defined as the need for at least 1 hemodialysis or doubling of pre-surgical creatinine levels), stroke and seizures (clinically diagnosed), myocardial infarction (new Q waves in two electrocardiogram leads), cardiac arrest, respiratory failure, re-operation and death. Monitoring of the patients prior to discharge involved chart review during their stay in the hospital; if a post-operative complication was suspected, the complication was confirmed using Montefiore Medical Center's Carecast Database, which contained independent results such as MRI's, CT scans, or labs. Additionally, computer records of the patients were searched to determine if there were documented complications in the 30-day post-operative time period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Subjects scheduled to undergo cardiac surgery requiring cardiopulmonary bypass

Exclusion Criteria:

* Vulnerable patient populations (unable to consent)
* Religious or other prohibitive reason for not receiving blood transfusion
* History of allergy to epsilon-aminocaproic acid or tranexamic acid
* Pregnant or breast-feeding (if applicable)
* The participation in another clinical or device trial that would affect the patient's coagulation profile
* Cardiac or cardiopulmonary transplantation procedure
* Any history of stroke and/or non-coronary thrombotic disorders (DVT, PE)
* Clinical signs consistent with non-coronary thrombotic disease
* Known congenital deficiency of Protein C, Protein S, Antithrombin and homozygous Factor V Leiden
* Known congenital bleeding disorders
* Weight < 50 kg
* Weight > 150 kg
* Acute renal failure or creatinine > 2.0 mg/dL
* Current surgery including any implantable ventricular assist device requiring CPB including ECMO (extracorpeal membrane oxygenation)
* Current surgery including the aortic arch and/or descending thoracic aorta
* Any changes to the planned surgery, which result int he patient not requiring CPB or meeting exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Leff, MD, Principal Investigator — Montefiore Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Started | 56 | 58
Completed | 56 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA) | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [54 to 76] | 65 [57 to 76] | 64 [56 to 76]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 19 | 28 | 47
  Male | 37 | 30 | 67
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56 | 58 | 114

OUTCOME MEASURES:

1. Primary Outcome: Chest Tube Drainage
Description: Chest tube drainage are collected from the nursing records, every 4th hourly the amount fluid collected is reported in the collection sheets.
Time Frame: 4 hours, 8 hours, 12 hours, 24 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
mL
  4 hr | 200 (375) | 225 (400)
  8 hr | 375 (550) | 400 (675)
  12 hr | 425 (750) | 500 (825)
  24 hr | 700 (1100) | 800 (1225)

2. Primary Outcome: Median Amount of Blood Products Used
Description: Four types of blood products may be given through blood transfusions: whole blood, red blood cells, platelets, and plasma
Time Frame: 24 hours after surgery
Measure: Median (Standard Deviation); unit: L
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
L | .59 (1.3) | 1.20 (2.2)

3. Secondary Outcome: Diagnosis of Renal Dysfunction Post-operation
Description: Confirmed diagnosis of renal dysfunction and hospitalization for the same within 30 days after the surgery
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 3 | 2

4. Secondary Outcome: Diagnosis of Myocardial Infarction Post-operation
Description: Confirmed diagnosis of myocardial infraction and hospitalization for the same within 30 days after the surgery
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Epsilon-aminocaproic Acid (EACA); Tranexamic Acid (TA): How many subjects had a myocardial infarction?
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 1 | 1

5. Secondary Outcome: Number of Participants Who Have Confirmed Diagnosis of Respiratory Arrest
Description: Confirmed diagnosis of respiratory arrest and hospitalization for the same within 30 days after the surgery
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 11 | 5

6. Secondary Outcome: Number of Participants With Confirmed Diagnosis of Stroke
Description: Confirmed diagnosis of stroke and hospitalization for the same within 30 days after the surgery
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 2 | 2

7. Secondary Outcome: Number of Participants With Confirmed Diagnosis of Seizure
Description: Confirmed diagnosis of seizure and hospitalization for the same within 30 days after the surgery
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 0 | 0

8. Secondary Outcome: Reoperation
Description: Confirmed diagnosis of reopeartion and hospitalization for the same within 30 days after the surgery
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Epsilon-aminocaproic Acid (EACA); Tranexamic Acid (TA): How many subjects were reoperated on?
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 3 | 4

9. Secondary Outcome: Mortality Within 30 Days Post-operation
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Groups:
- Epsilon-aminocaproic Acid (EACA); Tranexamic Acid (TA): How many subjects passed away?
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
Number analyzed (Participants) | 56 | 58
Participants | 1 | 1

10. Other Pre Specified Outcome: Patient Demographics
Description: Measurements taken as a composite. BMI, Sex, Age are to be determined to ensure that the subjects' characteristics were comparable between the Epsilon-aminocaproic Acid and Tranexamic Acid groups.
Time Frame: Baseline
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Type of Surgery
Time Frame: Intraoperative
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Intraoperative Characteristics
Description: Measurements are taken as a composite to determine that the subjects' characteristics are comparable between the Epsilon-aminocaproic Acid and Tranexamic Acid groups. Measurements include temperature, Heparin dose, protamine given, time of surgery, time of cardiopulmonary bypass, and aortic clamp time.
Time Frame: Intraoperative
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Epsilon-aminocaproic Acid (EACA) | Tranexamic Acid (TA)
All-Cause Mortality (participants affected / at risk) | 1/56 | 1/58
Serious Adverse Events (participants affected / at risk) | 20/56 | 14/58
Other Adverse Events (participants affected / at risk) | 0/56 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epsilon-aminocaproic Acid (EACA) (N=56) | Tranexamic Acid (TA) (N=58)
Death (Cardiac disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 2 | 2
Renal Dysfunction (Renal and urinary disorders) | 3 | 2
Reoperation within 24 hours (Surgical and medical procedures) | 3 | 4
Seizure (Nervous system disorders) | 0 | 0
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 11 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes